CLINICAL TRIAL: NCT04130919
Title: A Phase 2, Blinded, Randomized, Placebo-Controlled Study Evaluating the Efficacy and Safety of GS-4875 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Study to Evaluate the Efficacy and Safety of Tilpisertib in Adults With Moderately to Severely Active Ulcerative Colitis
Acronym: Falcon
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated the study since a new molecular entity was able to achieve greater target coverage
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-365-4237; 2019-001430-33 (EudraCT Number)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tilpisertib 300 mg (Experimental): Participants will receive blinded tilpisertib 300 mg for up to 10 weeks. An efficacy assessment will be performed at Week 10. Participants who achieve MCS response will continue on the blinded treatment for up to 50 weeks.
  Interventions: Drug: Tilpisertib
- Tilpisertib 100 mg (Experimental): Participants will receive blinded tilpisertib 100 mg for up to 10 weeks. An efficacy assessment will be performed at Week 10. Participants who achieve MCS response will continue on the blinded treatment for up to 50 weeks.
  Interventions: Drug: Tilpisertib
- Placebo (Placebo Comparator): Participants will receive blinded tilpisertib matching placebo for up to 10 weeks. An efficacy assessment will be performed at Week 10. Participants who achieve MCS response will continue on the blinded treatment for up to 50 weeks.
  Interventions: Drug: Placebo
- Open-label Tilpisertib 300 mg (Experimental): Based on the efficacy assessment results at Week 10, participants who do not achieve MCS response will have the option to receive open-label tilpisertib 300 mg for up to 50 weeks.
  Interventions: Drug: Tilpisertib

INTERVENTIONS:
Drug: Tilpisertib — Tablets administered orally once daily
  Other Names: GS-4875
  Arms: Open-label Tilpisertib 300 mg; Tilpisertib 100 mg; Tilpisertib 300 mg
Drug: Placebo — Tablets administered orally once daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of tilpisertib (formerly GS-4875) compared with placebo control in achieving clinical remission per modified Mayo Clinic Score (MCS) in adults with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Key Inclusion Criteria:

* Males, or non-pregnant, non-lactating females, at least 18 years of age based on the date of the screening visit.
* UC of at least 3 months duration before randomization confirmed by endoscopy and histology at any time in the past AND a minimum disease extent of 15 centimeter (cm) from the anal verge. Documentation of endoscopy and histology consistent with the diagnosis of UC must be available in the source documents prior to the initiation of screening.
* Moderately to severely active UC as determined during screening by a centrally read endoscopy score ≥ 2, a Rectal Bleeding subscore ≥ 1, a Stool Frequency subscore ≥ 1 and Physicians Global Assessment (PGA) of ≥ 2 as defined by the Mayo Clinic Score; total MCS must be between 6 and 12, inclusive.
* Previously demonstrated an inadequate response (primary non-response) or loss of response (secondary non-response) to a tumor necrosis factor-alpha (TNFα) inhibitor (ie, infliximab, adalimumab, golimumab, or biosimilars). The induction treatment regimen resulting in inadequate response or loss of response should have been in accordance with local prescribing information/guidelines or as outlined below.

  * Infliximab: 5 mg/kg at Weeks 0, 2, and 6
  * Adalimumab: 160 mg on Day 1 (given in 1 day or split over consecutive days), followed by 80 mg 2 weeks later (Day 15), 40 mg 2 weeks later (Day 29) and every 2 weeks thereafter until Day 57
  * Golimumab: 200 mg on Day 1 followed by 100 mg at Week 2
* May be receiving concomitant therapy for UC at the time of enrollment as specified in the protocol, provided the dose prescribed has been stable as indicated prior to randomization.
* Meet the following Tuberculosis (TB) screening criteria:

  * No evidence of active TB, latent TB, or inadequately treated TB as evidenced by 1 of the following:

    * A negative QuantiFERON test or equivalent assay reported by the central lab at screening or within 90 days prior to randomization date. OR
    * A history of fully treated active or latent TB according to local standard of care. Investigator must verify adequate previous anti-TB treatment and provide documentation; these individuals do not require QuantiFERON testing and eligibility must be approved by the sponsor prior to enrollment in the study. AND
    * A chest radiograph (views as per local guidelines with the report or films available for investigator review) taken at screening or within the 4 months prior to randomization without evidence of active or latent TB infection.
* Laboratory assessments at screening within the following parameters:

  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and total bilirubin ≤ 2 X upper limit of normal (ULN)
  * Estimated glomerular filtration rate (eGFR) ≥ 60 ml/min (1.0 mL/sec) as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Cystatin C formula as described in protocol.
  * Hemoglobin ≥ 8 g/dL (≥ 80 g/L)
  * Absolute neutrophil count (ANC) ≥ 1.5 × 10^3/μL (≥ 1.5 GI/L)
  * Platelets ≥ 100 × 10^3/μL (≥ 100 GI/L)
  * White blood cells (WBC) ≥ 3 × 10^3/μL (≥ 3 GI/L)
  * Absolute lymphocyte count ≥ 0.75 × 10^3/μL (≥ 0.75 GI/L)

Key Exclusion Criteria:

* Currently displaying clinical signs of acute severe colitis, fulminant colitis, or toxic megacolon.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (49):
- United States (23):
  - Gut P.C., dba Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Om Research LLC, Lancaster, California
  - United Medical Doctors, Murrieta, California
  - Alliance Clinical Research, Poway, California
  - Alliance Medical Research, Coral Springs, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - A Plus Research, Inc, Miami, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Kansas City Research Institute, Kansas City, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - Allied Digestive Disease Center, Cypress, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants, San Marcos, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Australia (4):
  - Coastal Digestive Health, Maroochydore, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Emeritus Research, Melbourne, Victoria
- Austria (2):
  - Medizinische Universität Innsbruck, Universitätsklinik für Innere Medizin I, Innsbruck
  - Medizinische Universitat Wien Klinik fur Innere Medizin III/Abt. fur Gastroenterologie and Hepatologie, Vienna
- Vancouver General Hospital - The Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada
- France (9):
  - Hopital Beaujon, Clichy
  - CHU de Dijon Bourgogne, Dijon
  - Centre Hospitalier Universitaire de Grenoble Alpes, Grenoble
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Lyon Sud, Pierre-Bénite
  - CHRU Pontchaillou, Rennes
  - CHU de Saint Etienne, Saint-Etienne
  - Hopital Rangueil, Toulouse
  - CHRU de Nancy, Vandœuvre-lès-Nancy
- Germany (3):
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik fur Innere Medizin I, Haus C, Haus K3, Kiel
  - Eugastro GmbH, Leipzig
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
- Istituto Clinico Humanitas, Rozzano, Italy
- Poland (3):
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - "GASTROMED" Kopon, Zmudzinski i Wsp. Sp. J. Spec. Centrum Gastrologii i Endoskopii, Spec. Gabinety Lekarskie, Torun
  - Centrum Medyczne Melita Medical, Wroclaw
- Switzerland (3):
  - Gastroenterologische Praxis Balsiger, Seibold & Partner/Crohn-Colitis-Zentrum, Bern
  - Inselspital Bern/Klinik fur Viszerale Chirurgie und Medizin/Bauchzentrum, Bern
  - Universitätsspital Zürich/Klinik für Gastroenterologie und Hepatologie, Zurich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe and the United States.
Pre-assignment Details: 32 participants were screened.
Groups:
- Tilpisertib 300 mg (Blinded Treatment Phase): Tilpisertib 300 mg tablet orally once daily up to Week 10. Participants who achieved clinical response per Modified Mayo Clinic score (MCS) at Week 10, continued to receive tilpisertib 300 mg tablets orally once daily for a maximum of 50 weeks in the Blinded Treatment phase.
- Tilpisertib 100 mg (Blinded Treatment Phase): Tilpisertib 100 mg tablet orally once daily up to Week 10. Participants who achieved clinical response per modified MCS at Week 10, continued to receive tilpisertib 100 mg tablets orally once daily for a maximum of 50 weeks in the Blinded Treatment phase.
- Placebo (Blinded Treatment Phase): Placebo tablet orally once daily up to Week 10. Participants who achieved clinical response per modified MCS at Week 10, continued to receive placebo tablets orally once daily for a maximum of 50 weeks in the Blinded Treatment phase.
- Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase): Participants who received tilpisertib 300 mg and did not achieve clinical response per modified MCS at Week 10 in the Blinded Treatment phase, received tilpisertib 300 mg tablets orally once daily for up to 50 weeks in the Open-label Treatment phase.
- Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase): Participants who received tilpisertib 100 mg and did not achieve clinical response per modified MCS at Week 10 in the Blinded Treatment phase, received tilpisertib 300 mg tablets orally once daily for up to 50 weeks in the Open-label Treatment phase.
- Tilpisertib 300 mg From Placebo (Open-label Treatment Phase): Participants who received placebo and did not achieve clinical response per modified MCS at Week 10 in the Blinded Treatment phase, received tilpisertib 300 mg tablets orally once daily for up to 50 weeks in the Open-label Treatment phase.
Period: Blinded Treatment Phase
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase)
Started | 7 | 6 | 6 | 0 | 0 | 0
Completed | 5 | 4 | 3 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Disease worsening | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Investigator's decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-label Treatment Phase
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase)
Started | 0 (Participants who completed the Blinded Treatment phase and did not achieve the clinical response per modified MCS at Week 10 entered in Open-label Treatment phase to receive tilpisertib 300 mg.) | 0 (Participants who completed the Blinded Treatment phase and did not achieve the clinical response per modified MCS at Week 10 entered in Open-label Treatment phase to receive tilpisertib 300 mg.) | 0 (Participants who completed the Blinded Treatment phase and did not achieve the clinical response per modified MCS at Week 10 entered in Open-label Treatment phase to receive tilpisertib 300 mg.) | 4 (Participants who completed the Blinded Treatment phase and did not achieve the clinical response per modified MCS at Week 10 entered in Open-label Treatment phase to receive tilpisertib 300 mg.) | 3 (Participants who completed the Blinded Treatment phase and did not achieve the clinical response per modified MCS at Week 10 entered in Open-label Treatment phase to receive tilpisertib 300 mg.) | 3 (Participants who completed the Blinded Treatment phase and did not achieve the clinical response per modified MCS at Week 10 entered in Open-label Treatment phase to receive tilpisertib 300 mg.)
Completed | 0 | 0 | 0 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 3 | 2 | 3
Not completed — Withdrew consent | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Disease worsening | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Investigator's decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — MCS response not achieved at open-label week 10 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Tilpisertib 300 mg (Blinded Treatment Phase): Tilpisertib 300 mg tablet orally once daily up to Week 10. Participants who achieved clinical response per modified MCS at Week 10, continued to receive tilpisertib 300 mg tablets orally once daily for a maximum of 50 weeks in the Blinded Treatment phase.
- Total: Total of all reporting groups
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase) | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.8) | 49 (22.6) | 43 (18.4) | 48 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 6
  Male | 5 | 5 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Race: Asian | 0 | 0 | 0 | 0
    Race: Black or African American | 0 | 0 | 2 | 2
    Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Race: White | 7 | 6 | 3 | 16
    Race: Other | 0 | 0 | 1 | 1
    Race: Not Permitted | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 6 | 4 | 6 | 16
    Ethnicity: Hispanic or Latino | 1 | 2 | 0 | 3
    Ethnicity: Not Permitted | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 1 | 0 | 1 | 2
  United States | 3 | 3 | 4 | 10
  Australia | 1 | 1 | 1 | 3
  Switzerland | 2 | 1 | 0 | 3
  Germany | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission Per Modified Mayo Clinic Score (MCS) at Week 10
Description: The modified MCS is a scoring system for assessment of ulcerative colitis (UC) activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal), and physician's global assessment (PGA) (range: 0 to 3, where 0 = normal and 3 = severe disease). Total score for MCS ranges from 0 to 12 (sum of all subscores), with higher scores indicating higher disease activity. Clinical remission per modified MCS is defined as stool frequency subscore ≤ 1 and not greater than baseline, rectal bleeding subscore of 0, and endoscopic subscore ≤ 1 at Week 10.
Time Frame: Week 10
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase)
Number analyzed (Participants) | 7 | 6 | 6
percentage of participants | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Who Achieved Endoscopic Response at Week 10
Description: Endoscopic response was defined as an endoscopic subscore of ≤ 1 at Week 10. Endoscopic subscore is a part of the modified MCS which is a scoring system for assessment of UC activity. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern), 2 = moderate disease (marked erythema, lack of vascular pattern, friability, erosions), and 3 = severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 10
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase)
Number analyzed (Participants) | 7 | 6 | 6
percentage of participants | 14.3 | 16.7 | 0

3. Secondary Outcome: Percentage of Participants Who Achieved MCS Response at Week 10
Description: The modified MCS is a scoring system for assessment of UC activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal), and PGA (range: 0 to 3, where 0 = normal and 3 = severe disease). Total score for MCS ranges from 0 to 12 (sum of all subscores), with higher scores indicating higher disease activity. MCS response is defined as a decrease from baseline of ≥ 3 points and at least 30% in MCS, in addition to a ≥ 1 point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore ≤ 1 at Week 10.
Time Frame: Week 10
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase)
Number analyzed (Participants) | 7 | 6 | 6
percentage of participants | 28.6 | 16.7 | 16.7

4. Secondary Outcome: Percentage of Participants Who Achieved MCS Remission at Week 10
Description: The modified MCS is a scoring system for assessment of UC activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal), and PGA (range: 0 to 3, where 0 = normal and 3 = severe disease). Total score for MCS ranges from 0 to 12 (sum of all subscores), with higher scores indicating higher disease activity. MCS remission is defined as a MCS score of ≤ 2 and no individual subscore > 1 at Week 10.
Time Frame: Week 10
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase)
Number analyzed (Participants) | 7 | 6 | 6
percentage of participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Achieved Histologic Remission Based Upon the Geboes Scale at Week 10
Description: Geboes histologic remission was assessed using the Geboes histologic scores to identify histologic changes in ulcerative colitis. Possible scores are Grade 0:Architectural changes(0.0=No abnormality to 0.3=Severe diffuse or multifocal abnormalities); Grade 1:Chronic inflammatory infiltrate(1.0=No increase to 1.3=Marked increase);Grade 2A:Eosinophils in lamina propria(2A.0=No increase to 2A.3-=Marked increase; Grade 2B:Neutrophils in lamina propria(2B.0= No increase to 2B.3=Marked increase);Grade 3:Neutrophils in epithelium (3.0=None to 3.3=>50% crypts involved);Grade 4:Crypt destruction(4.0=none to 4.3=Unequivocal crypt destruction),and Grade 5:Erosions and ulcerations:(5.0=No erosion, ulceration or granulation to 5.4=Ulcer or granulation tissue). Histologic remission defined as having Grade 0 of ≤ 0.3, Grade 1 of ≤ 1.1, Grade 2a of ≤ 2A.3, Grade 2b of 2B.0, Grade 3 of 3.0, Grade 4 of 4.0, and Grade 5 of 5.0. Geboes score ranges from 0 to 5.4. Lower values indicate better outcome.
Time Frame: Week 10
Population: Participants in the Full Analysis Set with at least 1 histological assessment were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase)
Number analyzed (Participants) | 6 | 6 | 4
percentage of participants | 16.7 | 16.7 | 25.0

6. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) for the Blinded Treatment phase are either defined as AEs with an onset date on or after the Blinded Treatment phase study drug start date and no later than 30 days after permanent discontinuation of the Blinded Treatment phase study drug if no Open-label Treatment phase study drug was taken, or any AEs with an onset date on or after the Blinded Treatment phase study drug start date and before the Open-label Treatment phase study drug start date if Open-label Treatment phase study drug was taken and/or any AEs leading to premature discontinuation of Blinded Treatment phase study drug. TEAEs for the Open-label Treatment phase are either defined as AEs with an onset date on or after the Open-label Treatment phase study drug start date and no later than 30 days after permanent discontinuation of the Open-lab Treatment phase study drug and/or any AEs leading to premature discontinuation of Open-label Treatment phase study drug.
Time Frame: Blinded Treatment phase: First dose date up to 50.6 weeks plus 30 days; Open-label phase: First dose date up to 50.7 weeks plus 30 days
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase)
Number analyzed (Participants) | 7 | 6 | 6 | 4 | 3 | 3
percentage of participants | 57.1 | 50.0 | 50.0 | 50.0 | 66.7 | 66.7

7. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities for Blinded Treatment phase are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of Blinded Treatment phase study drug plus 30 days for participants who permanently discontinued Blinded Treatment phase study drug or before the first dose of Open-label Treatment phase study drug. For the Open-label Treatment phase, treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from Open-label baseline at any postbaseline time point, up to and including the date of last dose of Open-label Treatment phase study drug plus 30 days for participants who permanently discontinued Open-label phase study drug. For maximum postbaseline toxicity grade, the most severe graded abnormality from all tests was counted for each patient. Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening.
Time Frame: as for outcome 6
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase)
Number analyzed (Participants) | 7 | 6 | 6 | 4 | 3 | 3
percentage of participants
  Grade 1 | 42.9 | 66.7 | 16.7 | 25.0 | 33.3 | 66.7
  Grade 2 | 28.6 | 33.3 | 50.0 | 25.0 | 0 | 33.3
  Grade 3 | 14.3 | 0 | 0 | 25.0 | 66.7 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: Blinded Treatment phase: First dose date up to 50.6 weeks plus 30 days; Open-label Treatment phase: First dose date up to 50.7 weeks plus 30 days; All-Cause Mortality: Enrollment up to Week 70.3
Description: Adverse Events: Safety Analysis Set included all participants who received at least one dose of study drug; All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
Arm/Group | Tilpisertib 300 mg (Blinded Treatment Phase) | Tilpisertib 100 mg (Blinded Treatment Phase) | Placebo (Blinded Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 1/6 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 4/7 | 3/6 | 2/6 | 2/4 | 2/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tilpisertib 300 mg (Blinded Treatment Phase) (N=7) | Tilpisertib 100 mg (Blinded Treatment Phase) (N=6) | Placebo (Blinded Treatment Phase) (N=6) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) (N=4) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) (N=3) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase) (N=3)
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tilpisertib 300 mg (Blinded Treatment Phase) (N=7) | Tilpisertib 100 mg (Blinded Treatment Phase) (N=6) | Placebo (Blinded Treatment Phase) (N=6) | Tilpisertib 300 mg From Tilpisertib 300 mg (Open-label Treatment Phase) (N=4) | Tilpisertib 300 mg From Tilpisertib 100 mg (Open-label Treatment Phase) (N=3) | Tilpisertib 300 mg From Placebo (Open-label Treatment Phase) (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Gilead made the decision to discontinue the development of tilpisertib since a new molecular entity was able to achieve greater target coverage. The decision was not due to any safety concerns. Since only 19 participants were enrolled, none of the planned statistical analyses were performed. During the coronavirus disease 2019 (COVID-19) pandemic, there were changes to protocol visits and procedures where necessary to mitigate the impact of the pandemic to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT04130919/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04130919/SAP_001.pdf